CLINICAL TRIAL: NCT04051528
Title: Do Combinatorial Training Lead to Better Cognition and Daily Participation in TBI Persons With Cognitive Impairments: Efficacy and Neural Mechanism of Combining Computerized Cognitive Training, Aerobic Exercise and Guided Training
Brief Title: Do Combinatorial Training Lead to Better Cognition and Daily Participation in TBI Persons With Cognitive Impairments
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 201802226B0A3
Record Dates: First submitted 2019-08-07; First posted 2019-08-09 (Actual); Last update posted 2021-06-21 (Actual); Status verified 2021-06

CONDITIONS: Trauma, Brain; Cognitive Deficit
Keywords: combinatorial training
MeSH Terms: conditions — Brain Injuries, Traumatic; Cognition Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- combinatorial training group (Experimental): Combinatorial training group will have the same procedure with the sequential training group in the first 8 sessions. After that the procedure for sessions from 9th to 16th will be 60 minutes of guiding training.
  Interventions: Procedure: aerobic exercise training; Procedure: computerized cognitive training; Procedure: guiding training
- sequential training group. (Experimental): Sequential training group will first undergo aerobic exercise training for 30 minutes followed by 30 minutes of computerized cognitive training. The difficult level of this training program will be adjusted automatically and continuously based on each participant's level of performance.
  Interventions: Procedure: aerobic exercise training; Procedure: computerized cognitive training

INTERVENTIONS:
Procedure: aerobic exercise training — The aerobic exercise will first perform 3 minutes of warm-up followed by 25 minutes of resistive aerobic exercise and then 2 minutes cool-down. During the aerobic exercise the target heart rate will be 40 to 70% of maximal heart rate calculated as (208 - 0.7 age). The exercise intensity will be progressed as the participants improve their performance throughout practice. Vital signs and the Borg Perceived Exertion Scale will be monitored and recorded during exercise for each session.
Procedure: computerized cognitive training — The core function of cognitive training will be including attention, recognition, color and shape identification, calculation, visual perception, visuospatial processing and executive function. Participants will perform tasks designed to enhance abovementioned types of cognitive functions. The difficult level of this training program will be adjusted automatically and continuously based on each participant's level of performance. Cognitive training group will use commercialized cognitive based training programs to facilitate several cognitive functions. The core function will be including attention, recognition, color and shape identification, calculation, visual perception, visuospatial processing and executive function. Participants will perform tasks designed to enhance abovementioned types of cognitive functions. The difficult level of this training program will be adjusted automatically and continuously based on each participant's level of performance.
Procedure: guiding training — At the first time in guiding training will focus on introducing the Goal-Plan-Do-Check strategy and identifying initial three goals by the Canadian Occupational Performance Measure. At the second time in guiding training will begin with a review of the Goal-Plan-Do-Check and will apply the Goal-Plan-Do-Check to the first initial goal. Participants will review this goal and plan, describe the execution of the plan (do), and evaluate the execution of the plan (check). After each execution of the plan, the participant will rate his performance using the COPM Performance Scale, producing iterative scores for each activity. The remaining session of guiding sessions will repeat this process, review performance of identified activities, and applying the Goal-Plan-Do-Check strategy to improve performance.
  Arms: combinatorial training group

SUMMARY:
The objectives of this study are to: (1) determine the effects of combinatorial training (i.e. combinatory of aerobic exercise with cognitive training and guiding training) vs. the sequential training (i.e. a combination of aerobatic exercise with cognitive training) on cognitive function, physical function, and daily function/participation and psychological function in persons with cognitive impairments post Traumatic brain injury (TBI); (2) determine the long-term effects of these two types of interventions on these outcome measures.

DETAILED DESCRIPTION:
Cognitive deficits and dysfunction in daily participation are common in patients with traumatic brain injury. Previous studies have reported positive effects on cognitive function after computerized cognitive training, aerobic exercise, or a combination of the two, however, the effects are variable and hardly be transferred to enhance daily participation. It is thus still inconclusive that which types of interventions are better for cognitive remediation and daily participation in patients post traumatic brain injury. Several pioneering studies used guided training for patients with brain injury to acquire problem-solving skills, improve life function and promote participation. After the training, the effect lasted for six months. However, due to insufficient research samples, it was inferior in generalizability.

In the present project, the investigators design an innovative combinatorial training that composites of guided training, computerized cognitive training, and aerobic exercise. The investigators expected that this combinatorial training not only improve cognitive ability but also facilitate daily participation in patients with traumatic brain injury. The investigators plan to recruit 50 patients with traumatic brain injury who have cognitive deficits and will assign them randomly into two groups: sequential training group, and combinatorial training group.

There will compare the immediate effects and long-term effects of combinatorial training and combined training (computerized cognitive training plus aerobic exercise) on cognitive function and daily function/participation and psychological function of persons with traumatic brain injury.

ELIGIBILITY:
Inclusion Criteria:

* (1) first episode non-progressive traumatic brain injury at least six months;
* (2) Age range from 18 to 65 years;
* (3) Rancho Los Amigo Level of Cognitive Functioning Scale (LOCF) = 7;
* (4) Montreal cognitive assessment (MOCA) < 26;
* (5) Self- or informant-reported memory or cognitive complaints;
* (6) Able to follow the study instruction;
* (7) Adequate cardiopulmonary function to perform aerobic exercise;
* (8) Able to walk with or without assistive devices.

Exclusion Criteria:

* (1) Unstable medical history (e.g., recent myocardial infarction) that might limit involving the training process;
* (2) Concomitant with other neurological disorders (e.g., Parkinson's disease, amyotrophic lateral sclerosis, multiple sclerosis);
* (3) Current participation in another interventional trial.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2020-06-03 (Actual); Primary Completion 2021-07 (Estimated); Study Completion 2022-01 (Estimated)

PRIMARY OUTCOMES:
Change scores of Montreal Cognitive Assessment (MoCA) | Baseline, post test immediately after completing 16 intervention sessions (around 8 weeks after baseline), follow up test (6 months after completing intervention sessions)
  The Montreal Cognitive Assessment (MoCA) will be used to assess general cognitive functions. It examines several cognitive domains with a total score of 30 and higher values indicate better cognitive functions. The MoCA has been shown to be a valid and promising tool to evaluate the global cognitive function in patients with stroke. The psychometric properties of MoCA are good to excellent for patients with cerebrovascular diseases.
Change scores of Wechsler Memory Scale - Third Edition (WMS-III) | Baseline, post test immediately after completing 16 intervention sessions (around 8 weeks after baseline), follow up test (6 months after completing intervention sessions)
  Several subtests of Wechsler Memory Scale - Third Edition (WMS-III) including Faces Recognition (total scale=48), Verbal Paired Associates (total scale = 32), Word Lists (total scale = 48), and Spatial Span (total scale=32) will be used to assess the immediate, delayed, and working memory tests. For each subtest, a higher number indicates better performance in memory function. The raw score of subtests will also be transferred to standardized Z scores and summed to represent an index of general memory function.
Change scores of Stroop Color-Word test | Baseline, post test immediately after completing 16 intervention sessions (around 8 weeks after baseline), follow up test (6 months after completing intervention sessions)
  The Stroop Color-Word test assesses the abilities of selective attention, inhibition and executive function. The participants will be tested under congruent and incongruent conditions. In the congruent condition, the participant will name the color ink of a word which is consistent with the written color name; whereas in the incongruent condition the participant will name the color ink differs from the written color name. In both conditions, the number of colors correctly named within 45 seconds will be measured and the performance in the congruent condition will be compared with the incongruent condition (Quaney et al., 2009).
Change scores of Trail Making Test (TMT) | Baseline, post test immediately after completing 16 intervention sessions (around 8 weeks after baseline), follow up test (6 months after completing intervention sessions)
  The TMT is a neuropsychological test of visual attention and task switching. It consists of two parts (TMT-A and TMT- B) in which the subject is instructed to connect a set of 25 dots as quickly as possible while still maintaining accuracy. The Chinese version of the TMT has been suggested to be a reliable instrument for measuring executive function among older adults. The scores for both TMT A and B are reported as the number of seconds required to complete the task. According to the TMT directions for administration, an average score for the TMT Part A is 29 seconds and a deficient score is greater than 78 seconds. For the TMT Part B, an average score is 75 seconds and a deficient score is greater than 273 seconds. Therefore, higher scores reveal greater impairment.
Change scores of Six-minutes Walking Test (6MWT) | Baseline, post test immediately after completing 16 intervention sessions (around 8 weeks after baseline), follow up test (6 months after completing intervention sessions)
  The 6MWT measures the maximum distance walked over 6 minutes, which assess the endurance and mobility level of the participants. The participants could rest as needed during the course of the test. The test-retest reliability and responsiveness has been established to be high for patients with chronic stroke (Fulk, Echternach, Nof, & O'Sullivan, 2008).
Change scores of 30-second Chair-Stand Test (30CST) | Baseline, post test immediately after completing 16 intervention sessions (around 8 weeks after baseline), follow up test (6 months after completing intervention sessions)
  The 30 second chair stand test (CST) will be assessed to indicate the strength and endurance level of the lower extremities. The participants will be asked to stand up from a standardized chair and then sit down as many times as possible within 30 seconds. The feasibility and reliability of using CST in people with cognitive impairment have been established to be good (Blankevoort et al., 2013).
Change scores of Berg Balance Scale (BBS) | Baseline, post test immediately after completing 16 intervention sessions (around 8 weeks after baseline), follow up test (6 months after completing intervention sessions)
  The Berg balance scale is a test of a person's static and dynamic balance abilities. This scale comprises a set of 14 simple balance related tasks, ranging from standing up from a sitting position, to standing on one foot. The degree of success in completing each task is given a score of zero (unable) to four (independent), and the final measure is the sum of all scores. The range of score is 0-56 and a below average score indicates a high risk for falls. Excellent test-retest reliability has been reported in acquired brain injury.
Change scores of Lower extremity muscle strength. | Baseline, post test immediately after completing 16 intervention sessions (around 8 weeks after baseline), follow up test (6 months after completing intervention sessions)
  We will evaluate isometric knee flexors and extensors muscle strength using handheld dynamometer. The participant will be seated upright in a chair with back support, the knee will be placed in 90-degree flexion and the evaluator will stabilize the thing to eliminate synergistic movements. Participants will be asked to perform a maximal isometric contraction of knee flexion and extension with affected and less affected side. We will record the mean value of 3 attempts.
Change scores of Mobility Level | Baseline, post test immediately after completing 16 intervention sessions (around 8 weeks after baseline), follow up test (6 months after completing intervention sessions)
  An objective measure of the amount of arm movements in real-life situations will be provided by the accelerometers. Actigraphy activity monitors (ActiGraph, Shalimar, FL, USA) will be worn on participants' wrists for 3 consecutive days before and after training to measure the number of moves each minute, and the average counts of move per minute. The participants will be asked to wear the device during the day and data recorded by the actigraphy will be analyzed with the MAHUFFE software (http://www.mrc-epid.cam.ac.uk/). The use of actigraphy has been validated for patients with TBI.
Change scores of Timed Up and Go test (TUG) | Baseline, post test immediately after completing 16 intervention sessions (around 8 weeks after baseline), follow up test (6 months after completing intervention sessions)
  The TUG assesses the dynamic balance ability and mobility. The participants will be required to stand up from a chair, walk 3 meters, turn around, walk back to the chair, and sit down. The test-retest reliability of TUG on individuals with stroke was excellent (Ng & Hui-Chan, 2005).
Change scores of Functional Independence Measure (FIM) | Baseline, post test immediately after completing 16 intervention sessions (around 8 weeks after baseline), follow up test (6 months after completing intervention sessions)
  The FIM assesses the dependence level of individuals with stroke to perform 18 activities (13 motor and five cognitive tasks) in daily living. The score ranges from 18 to 126 and higher scores demonstrate greater independent participation in daily activities (Ottenbacher, Hsu, Granger, & Fiedler, 1996). The FIM has good interrater reliability and validity (Hsueh, Lin, Jeng, & Hsieh, 2002).
Change scores of Activity Outcome Measurement for Post-Acute Care (AM-PAC) | Baseline, post test immediately after completing 16 intervention sessions (around 8 weeks after baseline), follow up test (6 months after completing intervention sessions)
  The AM-PAC assess difficulties in daily participation with 58 items containing the following aspects: physical functioning, self-care, daily routine, communication, and interpersonal interaction. The items and scoring system are adopted from the ICF framework. The AM-PAC has adequate reliability and validity. There are three specific functional domains: basic mobility(score range=18-72), daily activity(score range=15-60) and applied cognitive(score range=19-76). For each subtest, a higher score indicates better performance.
Change scores of Participation Measure-3 Domains, 4 Dimensions (PM-3D4D) | Baseline, post test immediately after completing 16 intervention sessions (around 8 weeks after baseline), follow up test (6 months after completing intervention sessions)
  The PM-3D4D includes 24 items measuring participation in productivity(6 items), social(12 items), and community(6 items) domains across 4 dimensions: diversity of participation(Y/N), frequency of participation(0-6), desire for change(Y/N), and difficulty in participation(1-4). The score of diversity of participation is percent of the number of items in which a person answered yes divided by the total number of items within each domain. The score of frequency of participation is sum of the ratings divided by the total number of items within each domain. The score of desire for change is percent of the number of items in which a person answered yes divided by the total number of items within each domain. The score of difficulty in participation is total score within each domain. The PM-3D4D has been shown adequate reliability and validity in rehabilitation patients.
Change scores of Goal Attainment Scaling (GAS) | Baseline, post test immediately after completing 16 intervention sessions (around 8 weeks after baseline), follow up test (6 months after completing intervention sessions)
  The GAS assesses the extent to which patient's individual goals are achieved in the course of intervention. The GAS has been shown responsive to the change in cognitive rehabilitation. It used to quantify the extent to which treatment goals were achieved. Individual goals were evaluated in a standardized way, using predefined levels of achievement based on current and expected performance. A 5-point Goal Attainment Scale was used: the baseline level (-2), partial achievement (-1), the expected level of achievement (0), small better than expected levels (1), remarkably better than expected levels(2).
Change scores of Beck depression inventory-version II (BDI-II) | Baseline, post test immediately after completing 16 intervention sessions (around 8 weeks after baseline), follow up test (6 months after completing intervention sessions)
  The Beck depression inventory is a self-report measure of depression severity. Excellent reliability and validity have been established in patients with TBI. The BDI-II contains 21 questions, each answer being scored on a scale value of 0 to 3. The range of score is 0-63 and higher total scores indicate more severe depression.

CONTACTS AND LOCATIONS:
Overall Officials: Ching-yi Wu, ScD, Principal Investigator — Chang Gung Memorial Hospital
Locations (1):
- Chang Gung Memorial Hospital, Taoyuan District, Taiwan

IPD SHARING:
Plan to Share IPD: No